CLINICAL TRIAL: NCT01634321
Title: The Phase 4 Clinical Trial to Evaluate the Efficacy and Safety of Luphere Depot Inj. 3.75mg(Leuprolide Acetate 3.75mg) in Patients With Precocious Puberty; A Single, Open, Multi-center, Prospective Study
Brief Title: The Clinical Trial to Evaluate the Efficacy and Safety of Luphere Depot Inj. 3.75mg(Leuprolide Acetate 3.75mg) in Patients With Precocious Puberty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_LP1M002P
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

ARMS (1):
- Luphere (Experimental)
  Interventions: Drug: Luphere depot 3.75mg(Leuprolide acetate 3.75mg)

INTERVENTIONS:
Drug: Luphere depot 3.75mg(Leuprolide acetate 3.75mg)

SUMMARY:
The purpose of this Clinical Trial was to Evaluate the Efficacy and Safety of Luphere Depot Inj. 3.75mg(Leuprolide acetate 3.75mg) in patients with precocious puberty.

ELIGIBILITY:
Inclusion Criteria:

* 4~8 years & tanner stage ≥ 2

Exclusion Criteria:

* Previous treatment with GnRH analog therapy

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
At 24 weeks, percentage of subjects with suppression of peak-stimulated Luteinizing Hormone (LH) concentrations | At 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University medical center, Soo-won, South Korea